CLINICAL TRIAL: NCT01882088
Title: Phase IV Non Comparative Study of the Impact of Dietary Fiber Deficiency Correction Using Mucofalk® on Clinical Features and Motor Function of the Esophagus in Patients With Non-erosive Gastroesophageal Reflux Disease
Brief Title: Phase IV Study of the Impact of Dietary Fibers on Symptoms and Esophageal Motility in Patients With Non-erosive GERD
Acronym: OGIG-130-1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Russian Academy of Medical Sciences (Other)
Collaborators: Dr. Falk Pharma GmbH (Industry)
Responsible Party: Principal Investigator, Vasily Isakov, MD, PhD, AGAF, Professor, Russian Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ION RAMS; RussianAMS-1 (Other: RussianAMS)
Record Dates: First submitted 2013-06-16; First posted 2013-06-20 (Estimated); Results first posted 2019-08-01 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-07

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: GERD; psyllium; Lower esophageal sphincter; Esophageal motility; Dietary fiber; Heartburn; gastroesophageal reflux; non-erosive gastroesophageal reflux disease
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn | interventions — Psyllium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mucofalk (Experimental): Mucofalk 15 g/day i.e. 5 g TID per os, 15-20 min before meal
  Interventions: Drug: Mucofalk

INTERVENTIONS:
Drug: Mucofalk — Mucofalk 15 g/day i.e. 5 g TID per os, 15-20 min before meal
  Other Names: Psyllium

SUMMARY:
Gastroesophageal reflux disease (GERD) is a chronic condition, which may significantly decrease patients' quality of life due to the typical symptoms - heartburn and regurgitation. These are caused by increasing number of transient lower esophageal sphincter relaxations, regularly recurring reflux of gastric content into oesophagus, acidification of the esophagus and consequent esophageal mucosa damage. In addition, an important role is played by the increase in production of hydrochloric acid in the stomach, the slowdown in the evacuation of the contents from the stomach and increase of gastric and intra-abdominal pressure. All of these factors may depend on the patient's diet.

Theoretical premises of the positive influence of including dietary fiber on the course of gastroesophageal reflux disease may be the fact that dietary fiber may absorb nitric oxide (NO) containing in food, which in turn has relaxing effects on the lower esophageal sphincter. In addition, fiber deficiency has been shown to be associated with increased chance of developing hiatal hernia, which is associated with greater risk of the disease manifestations. There is lack of data to confirm that dietary interventions like higher dietary fiber intake may lead to lower frequency of GERD symptoms and influence objective criteria (those, obtained during esophageal pH-impedance (here and further: pH - pondus hydrogenii, i.e. quantity of hydrogen, a scale to measure acidity of a solution) recording and high resolution esophageal manometry).

Mucofalk® is a drug of plant origin, consisting of a shell seeds of Plantago ovata (ispaghula, psyllium). High content of mucuses in the composition of psyllium seed allows it to include to group of soft food fibers, which has fundamental value for the appointment of a drug at a number of diseases, when, for example, the use of coarse food fibres not recommended or contraindicated.

Mucofalk is the registered medicinal (registration number of the Russian State register of medicines P N014176/01, registration date 14.07.2008, manufacturer: Lozan Pharma Gesellschaft mit beschränkter Haftung (GmbH), packager: Dr. Falk Pharma GmbH, Germany). Recommended dosage and administration: orally, adults and children over 12 years - 1 pack. 2-6 times a day. Before use, the contents of 1 packet poured in a glass, in which slowly poured with cold water (150 ml), stir and drink immediately. Then drink another glass of liquid.

DETAILED DESCRIPTION:
During the study 14-days screening period is provided to evaluate H.pylori and endoscopic status of the patient and to confirm the presence of dietary fiber deficiency (based on standard computerized dietary questionnaire). On the baseline physical examination, GERD-Q questionnaire, GERD symptom severity scale (by Likert), Bristol stool scale, high resolution esophageal manometry and 24-hours esophageal pH-impedance studies are to be provided. Since baseline, up to day 10 Mucofalk 15 g/day in three times a day (TID) regimen is to be given. All the patient will receive standardized menu. Repeat evaluation of symptoms, high resolution esophageal manometry and 24-hours esophageal pH-impedance are to be done at the day 10 of the study.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of non-erosive form of Gastroesophageal Reflux disease
* Dietary fiber deficiency by dietary questionnaire
* pathological gastroesophageal reflux by 24-hours esophageal pH-impedance examination
* willingness to participate (signed informed consent)

Exclusion Criteria:

* presence of esophageal mucosal damages (esophagitis) by endoscopic evaluation
* gastrointestinal surgery in anamnesis
* current pregnancy or breast-feeding
* known hypersensitivity to Mucofalk or its components

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vasily A Isakov, MD,PhD,AGAF, Study Chair — Fed. Research Center of Nutrition and Biotechnology, Gastroenterology&Hepatology; Sergey Morozov, MD, PhD, Principal Investigator — Fed. Research Center of Nutrition and Biotechnology, Gastroenterology&Hepatology
Locations (1):
- Research Institute of Nutrition of Russian Academy of Medical Sciences, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, results of the study could be shared
Supporting Information: Study Protocol, ICF, CSR
Time Frame: within 2 years after study completion
Access Criteria: Official regulatory institutions request, official request by researchers or researchers organizations
URL: http://ion.ru

REFERENCES:
- [Background] Ronkainen J, Aro P, Storskrubb T, Lind T, Bolling-Sternevald E, Junghard O, Talley NJ, Agreus L. Gastro-oesophageal reflux symptoms and health-related quality of life in the adult general population--the Kalixanda study. Aliment Pharmacol Ther. 2006 Jun 15;23(12):1725-33. doi: 10.1111/j.1365-2036.2006.02952.x. PMID 16817916
- [Background] Terry P, Lagergren J, Ye W, Wolk A, Nyren O. Inverse association between intake of cereal fiber and risk of gastric cardia cancer. Gastroenterology. 2001 Feb;120(2):387-91. doi: 10.1053/gast.2001.21171. PMID 11159879
- [Background] Burkitt DP, James PA. Low-residue diets and hiatus hernia. Lancet. 1973 Jul 21;2(7821):128-30. doi: 10.1016/s0140-6736(73)93067-5. No abstract available. PMID 4124047
- [Background] Nilsson M, Johnsen R, Ye W, Hveem K, Lagergren J. Lifestyle related risk factors in the aetiology of gastro-oesophageal reflux. Gut. 2004 Dec;53(12):1730-5. doi: 10.1136/gut.2004.043265. PMID 15542505
- [Background] El-Serag HB, Satia JA, Rabeneck L. Dietary intake and the risk of gastro-oesophageal reflux disease: a cross sectional study in volunteers. Gut. 2005 Jan;54(1):11-7. doi: 10.1136/gut.2004.040337. PMID 15591498
- [Background] Karamanolis G, Tack J. Nutrition and motility disorders. Best Pract Res Clin Gastroenterol. 2006;20(3):485-505. doi: 10.1016/j.bpg.2006.01.005. PMID 16782525
- See also: Dr. Falk Pharma Gmbh — http://www.drfalkpharma.ru/about_us.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 36 patients were enrolled. 1 patient withdrew informed consent before day 0, 1 excluded due to non-compliance, 1 could not tolerate oesophageal manometry, in 1 case there was no possibility to perform the manometry. Migration of the pH-impedance probe was found in two patients. The data of these mentioned 6 patients were excluded from the analysis
Period: Overall Study
Arm/Group | Mucofalk
Started | 35 (35 patients were provided with psyllium in 5.0 sachets, 3 sachets per day for 10 days)
Completed | 30
Not Completed | 5
Not completed — Intolerance of esophageal manometry | 1
Not completed — no possibility to place the catheter | 1
Not completed — Protocol Violation | 1
Not completed — inadequate pH-impedance tracings | 2

BASELINE CHARACTERISTICS:
Population: The shown data are from those patients who successfully completed the study and whose complete data were available for the final analysis
Arm/Group | Mucofalk
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.7 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Russia | 30
body mass index, kg/m^2 [Mean (Standard Deviation); unit: kg/m^2] | 36.7 (6.9)
weight, kg [Mean (Standard Deviation); unit: kg] | 82.5 (17.9)
smoking status (yes) [Count of Participants; unit: Participants] — Number of participants who answered "yes" to the question about smoking status
  Participants | 6
alcohol intake (yes) [Count of Participants; unit: Participants] — Number of the participants who drank alcohol
  Participants | 14
alcohol use (g/day) [Mean (Standard Deviation); unit: g/day] | 1.1 (1.7)
basal dietary fiber intake, g/day [Mean (Standard Deviation); unit: g/day] | 6.0 (2.3)
hiatal hernia presence [Count of Participants; unit: Participants] | 16
hiatal hernia size [Mean (Standard Deviation); unit: cm] — Population: out of those who had hiatal hernia
  cm
    number analyzed (Participants) | 16
    (all) | 0.9 (0.5)
stools per week, n [Mean (Standard Deviation); unit: stools per week] — number of stools per week
  stools per week | 7.0 (2.0)
Number of Gastroesophageal Refluxes [Mean (Standard Deviation); unit: refluxes a day] — Number of gastroesophageal refluxes registered with 24-hours esophageal pH-impedance tracing
  refluxes a day | 67.9 (17.7)
Acid exposure time [Mean (Standard Deviation); unit: Percent of time pH<4 per 24-hours period] — Percent of time when pH values at 5 cm above upper border of the lower esophageal sphincter were less than 4, on 24-hours oesophageal pH-impedance study. Acid exposure time (AET) is a commonly accepted term
  Percent of time pH<4 per 24-hours period | 5.6 (4.8)
Number of acid gastroesophageal refluxes [Mean (Standard Deviation); unit: acid refluxes per day] — Number of acid refluxes is measured by 24-hours oesophageal pH-impedance recordings. Reflux was considered as acid when oesophageal pH was less than 4 and the impedance revealed backward flow of the stomach content into the oesophagus.
  acid refluxes per day | 43.2 (14.7)
Number of patients experiencing heartburn during 7 days prior to baseline [Count of Participants; unit: Participants] — Presence of heartburn during 7 days prior to baseline was assessed with the use of a standardized questionnaire. This data was then compared to the data obtained at point EOT
  Participants | 28
minimal lower esophageal sphincter pressure at rest, mm Hg [Mean (Standard Deviation); unit: mm Hg] — Obtained during high resolution oesophageal manometry study at the baseline
  mm Hg | 22.0 (9.4)
Mean resting lower esophageal sphincter (LES) pressure after 10 water swallows [Mean (Standard Deviation); unit: mm Hg] — The data are obtained during high resolution oesophageal manometry study, this outcome is measured after 10 water swallows by 5 ml each. In this section baseline characteristics are shown
  mm Hg | 20.5 (9.5)
Minimal Resting Lower Esophageal Sphincter (LES) Pressure After 10 Water Swallows [Mean (Standard Deviation); unit: mm Hg] — The results were obtained with the use of high resolution oesophageal manometry. This parameter is based on measurements of the pressure during 10 water swallows by 5 ml water each. Normally it takes 10-20 minutes to perform this test. Here baseline characteristics are shown
  mm Hg | 14.1 (8.0)
Residual Lower Esophageal Sphincter Pressure [Mean (Standard Deviation); unit: mm Hg] — These data are obtained with the use of high resolution oesophageal manometry on the day before treatment was initiated
  mm Hg | 7.5 (6.1)
Mean Lower Esophageal Sphincter Pressure (at Rest) [Mean (Standard Deviation); unit: mm Hg] — This parameter is obtained with the use of high-resolution esophageal manometry performed on the Day 1 of psyllium intake
  mm Hg | 22.0 (9.4)

OUTCOME MEASURES:

1. Primary Outcome: Number of Gastroesophageal Refluxes
Description: Number of gastroesophageal refluxes registered with 24-hours esophageal pH-impedance on the 10th day of psyllium intake. Statistical data represent the results of the comparison of the data obtained on the day 10 of study (EOT) with the baseline characteristics provided in the specific section
Time Frame: End of Treatment, on day 10 of psyllium intake
Population: Thirty-six patients were enrolled, complete data from 30 were included in the final analysis.
Measure: Mean (Standard Deviation); unit: refluxes
Arm/Group | Mucofalk
Number analyzed (Participants) | 30
refluxes | 42.4 (13.5)
Statistical Analysis 1: Comparison: Mucofalk; Data were analyzed using Statistica 10 software. Wilcoxon matched pairs test of non-parametric module was used to assess changes of the studied parameters after the course of fiber supplementation in comparison to baseline. A P value of 0.05 was considered statistically significant. Sample size calculation was performed using 1-Way ANOVA. Effect size calculation was performed for every comparison; Test type: Equivalence — Data were analyzed using Statistica 10 software. Wilcoxon matched pairs test of non-parametric module was used to assess changes of the studied parameters after the course of fiber supplementation in comparison to baseline. A P value of 0.05 was considered statistically significant. Sample size calculation was performed using 1-Way ANOVA. Effect size calculation was performed for every comparison; p = 0.000002, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Acid Exposure Time
Description: Percent of time with pH less than 4 at 5 cm above upper border of lower oesophageal sphincter per 24-hours oesophageal pH-impedance recording on the day 10 of psyllium intake. This outcome measure was compared to the baseline characteristics provided in the specific section of the study description
Time Frame: End of Treatment, on day 10 of psyllium intake
Population: Thirty-six patients were enrolled, complete data from 30 were included in the final analysis.
Measure: Mean (Standard Deviation); unit: Percent of time pH<4 per 24-hours period
Arm/Group | Mucofalk
Number analyzed (Participants) | 30
Percent of time pH<4 per 24-hours period | 5.5 (7.57)
Statistical Analysis 1: Comparison: Mucofalk; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.2, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Number of Acid Gastroesophageal Refluxes
Description: Number of acid refluxes was measured by 24-hours oesophageal pH-impedance recordings. Reflux was considered as acid when oesophageal pH was less than 4 and the impedance revealed backward flow of the stomach content into the oesophagus. Outcome measure reflects the data of day 10 of psyllium intake. Statistics reflects comparison between EOT and baseline data.
Time Frame: End of Treatment, on day 10 of psyllium intake
Population: 36 subjects were enrolled, data of 30 of them were included to the final analysis
Measure: Mean (Standard Deviation); unit: acid refluxes
Arm/Group | Mucofalk
Number analyzed (Participants) | 30
acid refluxes | 30.3 (15.3)
Statistical Analysis 1: Comparison: Mucofalk; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.002415, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Number of Patients Experiencing Heartburn During 7 Days Prior the Day 10 of Psyllium Intake
Description: Presence of heartburn during 7 days prior to the day 10 of psyllium intake was evaluated with a standardized questionnaire. This result was assessed at EOT
Time Frame: 7 days prior to EOT
Population: 36 patients were enrolled, data of 30 of them were included to the final analysis
Measure: Number; unit: Number of participants
Arm/Group | Mucofalk
Number analyzed (Participants) | 30
Number of participants | 12
Statistical Analysis 1: Comparison: Mucofalk; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.000438, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Minimal Lower Esophageal Sphincter Pressure at Rest
Description: Obtained during esophageal high resolution manometry study. End of treatment data were compared to the baseline. Per standard, resting pressure is measured during 30 seconds. High resolution manometry data on day 10 was compared to baseline.
Time Frame: End of Treatment, on day 10 of psyllium intake
Population: 36 patients were enrolled. data of the 30 of them were available for the final analysis
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Mucofalk
Number analyzed (Participants) | 30
mm Hg | 11.3 (9.4)
Statistical Analysis 1: Comparison: Mucofalk; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.023, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Mean Resting Lower Esophageal Sphincter (LES) Pressure After 10 Water Swallows at the End of Treatment (the Day 10 of Psyllium Intake)
Description: The data are obtained during high resolution esophageal manometry study on the day 10 of psyllium intake. This outcome is measured after 10 water swallows by 5 ml each. The study usually lasts for about 15 to 20 minutes. Data of high-resolution esophageal manometry examination at baseline and on the day 10 of psyllium intake were compared.
Time Frame: End of Treatment, on day 10 of psyllium intake
Population: 36 patients enrolled, data of the 30 of them were available for the final analysis
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Mucofalk
Number analyzed (Participants) | 30
mm Hg | 22.0 (10.3)
Statistical Analysis 1: Comparison: Mucofalk; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.11, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Minimal Resting Lower Esophageal Sphincter (LES) Pressure After 10 Water Swallows
Description: The results obtained during high resolution esophageal manometry studies. This parameter is obtained after 10 water swallows by 5 ml each. Data of high resolution esophageal manometry (examination usually lasts for 10-20 min) on the day 10 of psyllium intake were compared to the baseline characteristics. The data were compared to baseline characteristics
Time Frame: End of Treatment, on day 10 of psyllium intake
Population: 36 patients were enrolled, data of 30 of them were available for the final analysis
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Mucofalk
Number analyzed (Participants) | 30
mm Hg | 14.9 (6.4)
Statistical Analysis 1: Comparison: Mucofalk; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.008, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Residual Lower Esophageal Sphincter Pressure
Description: These data are obtained during high resolution esophageal manometry studies. The end of treatment characteristics were compared to the baseline ones.
Time Frame: End of Treatment, on day 10 of psyllium intake
Population: 36 non-erosive reflux disease (NERD) patients were enrolled, the data of 30 of them were available for the final analysis
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Mucofalk
Number analyzed (Participants) | 30
mm Hg | 7.0 (5.4)
Statistical Analysis 1: Comparison: Mucofalk; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.94, Wilcoxon (Mann-Whitney)

9. Other Pre Specified Outcome: Mean Lower Esophageal Sphincter Pressure (at Rest)
Description: This parameter is obtained with the use of high-resolution esophageal manometry performed on the Day 10 of psyllium intake.
Time Frame: End of Treatment, on day 10 of psyllium intake
Population: 36 subjects were enrolled, data of 30 of them were available for the final analysis
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Mucofalk
Number analyzed (Participants) | 30
mm Hg | 26.5 (11.3)
Statistical Analysis 1: Comparison: Mucofalk; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.37, Wilcoxon (Mann-Whitney)

10. Other Pre Specified Outcome: Stools Per Week
Description: Episodes of stools were calculated during 7-day period. Mean number at the end point was compared to the baseline one
Time Frame: 7 days
Population: 36 patients were enrolled, complete data of 30 of them were available for the final analysis
Measure: Mean (Standard Deviation); unit: stools per week
Arm/Group | Mucofalk
Number analyzed (Participants) | 30
stools per week | 8.0 (3.0)
Statistical Analysis 1: Comparison: Mucofalk; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.00002, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Mandatory individual (each subject) time point for the assessment of adverse events presence was the Day10 of psyllium intake (end of treatment). Each participant was asked to contact study team immediately in case of any adverse event and was provided with primary and backup telephone contacts including those to use outside the working hours.
Description: Standard definitions were used
Arm/Group | Mucofalk
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 0/35

LIMITATIONS AND CAVEATS:
Absence of placebo control. Due to the nature of psyllium and its preparation, it is almost impossible to produce a comparator of similar viscosity, solubility in water, and taste. Relatively small group of patients

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No